CLINICAL TRIAL: NCT04425954
Title: Early Retinal Vascular Modifications After Endoscopic Endonasal Pituitary Surgery: The Role of OCT- Angiography
Brief Title: Evaluation of Early Retinal Vascular Modifications After Endoscopic Endonasal Pituitary Surgery
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: PT 2006/20
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Endonasal Pituitary Surgery — Surgical treatment consisted of an endoscopic endonasal approach using a rigid 0-degree endoscope, 18 cm in length and 4 mm in diameter.

SUMMARY:
This study evaluates the retinal vascular features using optical coherence tomography angiography in patients that received endoscopic endonasal approach for the removal of an intra-suprasellar pituitary adenoma compressing the optic nerve.

DETAILED DESCRIPTION:
To investigate the potential role of optical coherence tomography angiography in predicting the postoperative recovery of retinal vascular network of the optic disc in patients before and at 3 months after Endoscopic Endonasal Approach for the removal of an intra-suprasellar pituitary adenoma compressing the optic nerve.

The optical coherence tomography angiography represents a novel and non-invasive diagnostic technique that allows a detailed analysis of retinal vascular features.

ELIGIBILITY:
Inclusion Criteria:

* age older than 45 years
* diagnosis of pituitary adenoma
* treatment-naïve with Endoscopic Endonasal Pituitary Surgery
* absence of other neurological diseases
* absence of vitreoretinal and vascular retinal diseases

Exclusion Criteria:

* age younger than 45 years
* No diagnosis of pituitary adenoma
* previous treatments with Endoscopic Endonasal Pituitary Surgery
* presence of neurological diseases
* presence of vitreoretinal and vascular retinal diseases

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 45 years with pituitary adenoma. They did not present other ophthalmological and neurological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Study of vessel density of the optic disc in patients underwent Endoscopic Endonasal Pituitary Surgery for the removal of an intra-suprasellar pituitary adenoma compressing the optic nerve. | 48 hours
  To evaluate the role of optical coherence tomography angiography in predicting the recovery of the vessel density of the optic disc after surgery, using optical coherence tomography angiography (OCTA). The parameter analyzed by OCTA was the vessel density of the optic disc (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy